CLINICAL TRIAL: NCT03587883
Title: Daily Intake of Cocoa Flavanols and Arterial Stiffness in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 547762
Record Dates: First submitted 2018-05-03; First posted 2018-07-16 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: flavanol; cocoa flavanols; arterial stiffness; blood pressure; step test

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked and cross-over dietary intervention study in healthy adults.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocoa Flavanol intervention (Experimental): Capsules containing Mars Cocoa Extract manufactured by the Cocoapro® process, providing 300 mg of cocoa flavanols per capsule: 900 mg of cocoa flavanols consumed daily for 2 weeks; 2 intervention periods: Cocoa flavanols I and cocoa flavanols II.
  Interventions: Other: Cocoa flavanols I; Other: Cocoa flavanols II
- Control intervention (Placebo Comparator): Cocoa-based, flavanol-free, control-matched capsules consumed for 2 weeks; 2 intervention periods: control I and control II.
  Interventions: Other: Control I; Other: Control II

INTERVENTIONS:
Other: Cocoa flavanols I — Capsules containing Mars Cocoa Extract manufactured by the Cocoapro® process and containing 300mg of cocoa flavanols per capsule consumed for 2 weeks.
  Arms: Cocoa Flavanol intervention
Other: Control I — Cocoa-based, flavanol-free, control-matched capsules consumed for 2 weeks.
  Arms: Control intervention
Other: Cocoa flavanols II — Capsules containing Mars Cocoa Extract manufactured by the Cocoapro® process and containing 300mg of cocoa flavanols per capsule consumed for 2 weeks.
  Arms: Cocoa Flavanol intervention
Other: Control II — Cocoa-based, flavanol-free, control-matched capsules consumed for 2 weeks.
  Arms: Control intervention

SUMMARY:
A randomized, double-masked and cross-over dietary intervention study to investigate the effects of diet supplementation with cocoa flavanols on arterial stiffness in healthy adult human subjects.

DETAILED DESCRIPTION:
Cocoa flavanols (CF) are plant-derived compounds commonly present in the human diet. Examples of flavanol-containing foods and beverages are apples, chocolate, tea, wine, berries, pomegranate and nuts. Flavanols encompass a group of different compounds, and the final profile of flavanols in foods will depend on multiple factors including plant origin, time of harvesting, storage, food processing, and cooking techniques. The term "cocoa flavanols" (CF) as used here refers to the particular profile of flavanols and procyanidins naturally found in cocoa beans, and CF mainly consist of the monomeric flavanol (-)-epicatechin and its oligomeric derivatives (procyanidins) containing up to 10 monomer subunits.

Accumulating data resulting from dietary intervention studies suggest that the intake of diets rich in flavanols can exert a beneficial cardiovascular health effect in humans. However, most of these investigations have been conducted with patients with diverse health complications (e.g. hypertension, diabetes and coronary heart disease) rather than healthy subjects. Thus, the interpretation of these data in the context of nutrition, primary prevention, and dietary recommendations is limited. In the current study, the investigators propose to investigate the effects of cocoa flavanol intake on arterial stiffness in a healthy population of adults. The investigators submit that this investigation will provide novel insights into the potential health benefits of dietary flavanols and procyanidins in the context of cardiovascular health in humans. The data resulting from this study will be key to the design of larger scale studies in this context, which are needed to comprehensively study the role of dietary flavanols and procyanidins with regard to potential dietary recommendations and public health.

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years old
* BMI 18.5 - 34.9 kg/m2
* Weight ≥ 110 pounds
* Previously consumed cocoa and peanut products, with no adverse reactions
* Having completed physical exercise similar to 5 MET within the last 2 months without having any physical limitations [e.g. i) Brisk walking (at 4 mph); ii) Mowing lawn; iii) Bicycling-light effort (10 mph) and iv) Playing tennis-doubles.]

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Non-English speaking*
* BMI ≥ 35 kg/m2
* More than 150 minutes of moderate-intensity aerobic activity or 75 minutes of vigorous-intensity aerobic activity weekly and more than two days a week of muscle strengthening activities that work all major muscle groups (CDC recommended physical activity guidelines for adults)
* Allergies to nuts, cocoa and chocolate products
* Active avoidance of coffee and caffeinated soft drinks
* A history of cardiovascular disease, stroke, renal, hepatic, or thyroid disease
* History of clinically significant depression, anxiety or other psychiatric condition
* History of difficult blood draws
* History of Raynaud's disease
* Indications of substance or alcohol abuse within the last 3 years
* Current use of herbal, plant or botanical supplements (multi-vitamin/mineral supplements are allowed)
* Blood Pressure >140/90 mm Hg
* Blood Pressure < 100/60 mm Hg, or heart rate < 50 bpm (due to limitations in the assessment of arterial stiffness
* GI tract disorders, previous GI surgery (except appendectomy)
* Self-reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food, potentially leading to bloating, cramping or gas)
* Diarrhea within the last month, or antibiotic intake within the last month
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, on a weight loss diet or individuals following diets with significant deviations from the average diet
* Metabolic panel results or complete blood counts that are outside of the normal reference range and are considered clinically relevant by the study physician
* Cold, flu, or upper respiratory condition at screening
* Currently participating in a clinical or dietary intervention study
* *Non-English speaking volunteers will be excluded for safety reasons, as we do not have staff that can adequately provide interpretation services that can explain and answer questions with regard to study procedures.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Individual changes in systolic blood pressure (in office) | Baseline and 2, 4, 6, 8 and 10 weeks following intervention
  assessed as systolic blood pressure
Individual changes in diastolic blood pressure (in office) | Baseline and 2, 4, 6, 8 and 10 weeks following intervention
  assessed as diastolic blood pressure
Individual changes in augmentation index (in office) | Baseline and 2, 4, 6, 8 and 10 weeks following intervention
  assessed as augmentation index
Individual changes in central blood pressure (in office) | Baseline and 2, 4, 6, 8 and 10 weeks following intervention
  assessed as central blood pressure
Individual changes in blood pressure (at home) | Daily for 2 weeks between 0, 2, 4, 6, 8 and 10 weeks of intervention
  self monitoring blood pressure
Individual changes in pulse wave velocity (in office) | Baseline and 2, 4, 6, 8 and 10 weeks following intervention
  assessed as pulse wave velocity
Individual changes in lipid profile | Baseline and 2, 4, 6, 8 and 10 weeks following intervention
  Total cholesterol, LDL, HDL and Triglycerides

SECONDARY OUTCOMES:
Individual changes in flavanol metabolites in plasma and urine | Baseline and 2, 4, 6, 8, 10 weeks following intervention
  flavanol/methylxanthine metabolites in plasma and urine
Individual changes in methylxanthine metabolites in plasma and urine | Baseline and 2, 4, 6, 8, 10 weeks following intervention
  flavanol/methylxanthine metabolites in plasma and urine
Individual changes in CMP | Baseline and 2, 4, 6, 8, 10 weeks following intervention
  comprehensive metabolic panel
Individual changes in Step test performance | Baseline and 2, 4, 6, 8, 10 weeks following intervention
  Volunteers will be asked to step up and down on a platform (7 inches high) at a rate of 23 steps per minute for no more than 3 minutes. Blood pressure will be measured before and after the step test.

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — UC Davis; Javier I Ottaviani, PhD, Study Director — Mars, Inc.
Locations (1):
- Ragle Human Nutrition Research Center, Department of Nutrition at UC Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schroeter H, Heiss C, Spencer JP, Keen CL, Lupton JR, Schmitz HH. Recommending flavanols and procyanidins for cardiovascular health: current knowledge and future needs. Mol Aspects Med. 2010 Dec;31(6):546-57. doi: 10.1016/j.mam.2010.09.008. Epub 2010 Sep 18. PMID 20854838